CLINICAL TRIAL: NCT01389362
Title: The Healing Effect of a Two-Herb Recipe on Foot Ulcer in Chinese Patients With Type 2 Diabetes: A Randomized, Placebo-Controlled Study
Brief Title: The Healing Effect of a Two-Herb Recipe on Foot Ulcer in Chinese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Prof. Chan Chung Ngor, Juliana, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRE-2008.581
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; foot ulcer; Chinese herbal medicine
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — rehmannia root; Huang Qi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese Herbal Medicine (Active Comparator): 2 sachets of Chinese Herbal Medicine to be taken daily
  Interventions: Drug: Chinese herbal medicine (Radix Rehmanniae and Radix Astragali)
- Placebo arm (Placebo Comparator): 2 sachets to be taken daily
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Chinese herbal medicine (Radix Rehmanniae and Radix Astragali) — 2 sachets to be taken daily
  Arms: Chinese Herbal Medicine
Drug: Placebo comparator — 2 sachets to be taken daily
  Arms: Placebo arm

SUMMARY:
There is now a global epidemic of diabetes and obesity affecting more than 300 million people worldwide with Asia in the forefront. In Hong Kong, diabetes affects more than 10% of the population. Patients with diabetes have a 12-25% lifetime risk of developing a foot ulcer.The abnormal metabolic milieus of hyperglycemia, hyperlipidemia, hypertension, pro-thrombotic state and chronic inflammation in diabetes causes atherosclerosis.A significant proportion of subjects have underlying peripheral arterial disease and neuropathy. These subjects are at great risk of developing infective foot ulceration secondary to impaired vascular supply, sensory loss and minor trauma.Without prompt and proper medical treatment, these infective ulcers will deteriorate leading to gangrene and limb amputation. In-vitro and in-vivo studies revealed that 5 out of the 12 herbs were effective in promoting fibroblast proliferation and angiogenesis. To minimize potential drug interactions and adverse effects from multiple components in a recipe of Traditional Chinese Medicine (TCM), the investigators have developed a simplified formula from the 12 herbs consisting of only two herbs. In this proof-of-concept study, the investigators hypothesize that the novel recipe of herbal medicine will expedite healing of early foot ulcer by promoting vascularisation and granulation as well as modulating inflammatory response.

DETAILED DESCRIPTION:
There is now a global epidemic of diabetes and obesity affecting more than 300 million people worldwide with Asia in the forefront. In Hong Kong, diabetes affects more than 10% of the population. Patients with diabetes have a 12-25% lifetime risk of developing a foot ulcer. These silent conditions independently and collectively contribute to 50% of all causes of death mainly due to cardiovascular and renal complications. Type 2 diabetes is a complex disorder characterized by a constellation of cardiovascular risk factors, notably, hyperglycemia, obesity, dyslipidemia (high triglyceride (TG) and low HDL-C), hypertension, microinflammation and prothrombotic state, often referred to as the metabolic syndrome. The public health implication of diabetes lies mainly in its devastating chronic complications due to generalized vascular dysfunction. In patients with diabetes and metabolic syndrome, loss of cellular structure or function due to apoptosis, angiogenesis and fibrosis eventually manifest as overt diabetic complications, such as cardiovascular diseases, neuropathy, retinopathy and nephropathy.

The abnormal metabolic milieus of hyperglycemia, hyperlipidemia, hypertension, pro-thrombotic state and chronic inflammation in diabetes causes atherosclerosis. A significant proportion of subjects have underlying peripheral arterial disease and neuropathy. These subjects are at great risk of developing infective foot ulceration secondary to impaired vascular supply, sensory loss and minor trauma. Without prompt and proper medical treatment, these infective ulcers will deteriorate leading to gangrene and limb amputation. Age, wound depth, the presence of ischaemia, a low albumin level, and the lack of simultaneous ulceration are the most significant independent predictors of an unfavourable outcome. The conventional management of diabetic foot ulcer includes rest, antibiotic therapy, surgical debridement and good glycemic control. The investigators previously demonstrated that the use of a recipe containing 12 herbs was effective in promoting the healing of severe chronic non-healing diabetic foot ulcers and achieved an 85% of limb preservation. In-vitro and in-vivo studies revealed that 5 out of the 12 herbs were effective in promoting fibroblast proliferation and angiogenesis. To minimize potential drug interactions and adverse effects from multiple components in a recipe of Traditional Chinese Medicine (TCM), the investigators have developed a simplified formula from the 12 herbs consisting of only two herbs.

Many herbs have long been used to treat diabetes mellitus and its complications. In many of these successful attempts Radix Rehmanniae (RR) and Radix Astragali (RA) have frequently been used in combination with other herbs to form complex formulae such as 'blood-house blood stasis-dispelling decoction with additive ingredients' and 'pills of six drugs with Rehmannia'.

Based on our previous in-vitro and in-vivo studies, a new reformulated recipe of herbal medicine has been developed. In this proof-of-concept study, the investigators hypothesize that the novel recipe of herbal medicine will expedite healing of early foot ulcer by promoting vascularisation and granulation as well as modulating inflammatory response. Results will provide valuable insight and understanding of the application of TCM in the management of diabetic foot ulcer, in particular, the effect on angiogenesis and anti-inflammation. New intellectual properties will be developed and provide the foundation for future research. Such an integrated approach from bench to bedside will serve as a model platform for the development of TCM in Hong Kong.

The study will investigate whether the two-herb recipe can increase the wound healing of patients with diabetes mellitus.

Primary outcome:

1. Resolution/progression of foot ulcer based on PEDIS
2. Failure of treatment i.e. no improvement in 6 months, rapid deterioration or emergency surgery required

Secondary outcome:

1. Hospital admission/attendance/stay
2. Metabolic parameters

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetic subjects with documented evidence of mild diabetic foot ulcer

* Male or female patients attending Diabetic Clinics and/or Podiatry Clinics at the hospitals of the New Territories East Cluster
* Aged between 20 and 75 years old inclusive
* All patients should be on stable dose of medication 4 weeks prior to enrolment
* Written informed consent
* If the patient is a woman of child-bearing potential, she must agree to use adequate method of contraception throughout the study period, unless surgically sterilized.

Exclusion Criteria:

Patients with end-stage renal disease as defined by the need for dialysis or on renal replacement program

* Patients with advanced diabetic eye disease as defined by the history of laser therapy, retinal detachment or vitreous hemorrhage
* Pregnancy, breast feeding, or patient has plans of becoming pregnant during the study period.
* Known allergy to TCM drugs
* Contraindication or intolerance to use of aspirin, statin , ACEI or ARB
* History of major gastrointestinal bleeding in the 5 years prior to consent
* Congestive heart failure of any severity
* Significant cardiovascular disease within 3 months of enrolment including acute coronary syndrome, cardiac revascularization procedure, transient ischemic attack and cerebrovascular accident
* HbA1c ≥ 10%
* Severe liver function impairment (≥ 3 ULN of ALT) and renal impairment (eGFR < 30 ml/min/1.73 m2)
* Investigational drugs within 30 days of enrolment
* Patient taking any Chinese herbal medicine in the 8 weeks prior to enrolment into the study
* Any other medical conditions that is considered as unsuitable for the study by investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Resolution/progression of foot ulcer based on PEDIS | 6 months

SECONDARY OUTCOMES:
Hospital admission/attendance/stay | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Juliana NA Chan, MBChB, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Diabetes and Endocrine Centre, Hong Kong SAR, Hong Kong SAR, China

REFERENCES:
- [Derived] Ko CH, Yi S, Ozaki R, Cochrane H, Chung H, Lau W, Koon CM, Hoi SW, Lo W, Cheng KF, Lau CB, Chan WY, Leung PC, Chan JC. Healing effect of a two-herb recipe (NF3) on foot ulcers in Chinese patients with diabetes: a randomized double-blind placebo-controlled study. J Diabetes. 2014 Jul;6(4):323-34. doi: 10.1111/1753-0407.12117. Epub 2014 Feb 24. PMID 24330156